CLINICAL TRIAL: NCT04402489
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate Efficacy, Safety, and Tolerability of MT-7117 in Adults and Adolescents With Erythropoietic Protoporphyria or X-Linked Protoporphyria
Brief Title: Study to Evaluate Efficacy, Safety, and Tolerability of MT-7117 in Subjects With Erythropoietic Protoporphyria or X-Linked Protoporphyria
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tanabe Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MT-7117-G01; jRCT2080225355 (Registry Identifier: Japan Registry of Clinical Trials (jRCT)); 2019-004226-16 (EudraCT Number)
Record Dates: First submitted 2020-05-20; First posted 2020-05-26 (Actual); Results first posted 2025-03-21 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: EPP; XLP

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo Comparator (Placebo Comparator): Oral tablet of placebo once a day.
  Interventions: Drug: Placebo
- MT-7117 Low Dose (Experimental): Oral tablet of MT-7117 Low Dose once a day.
  Interventions: Drug: MT-7117 Low Dose
- MT-7117 High Dose (Experimental): Oral tablet of MT-7117 High Dose once a day.
  Interventions: Drug: MT-7117 High Dose

INTERVENTIONS:
Drug: Placebo — Placebo
  Arms: Placebo Comparator
Drug: MT-7117 Low Dose — MT-7117 Low Dose
  Other Names: Dersimelagon
  Arms: MT-7117 Low Dose
Drug: MT-7117 High Dose — MT-7117 High Dose
  Other Names: Dersimelagon
  Arms: MT-7117 High Dose

SUMMARY:
The primary objective of this study is to investigate the efficacy of MT-7117 on time to onset and severity of first prodromal symptoms (burning, tingling, itching, or stinging) associated with sunlight exposure in adults and adolescents with EPP or XLP aged 12-75.

ELIGIBILITY:
Additional screening criteria check may apply for qualification.

Inclusion Criteria:

1. Subjects provided written informed consent to participate. For minor subjects, both minor assent and parental consent will be provided.
2. Male and female subjects with a confirmed diagnosis of EPP or XLP based on medical history, aged 12 years to 75 years, inclusive, at Screening.
3. Subjects have a body weight of ≥30 kg.
4. Subjects are willing and able to travel to the study sites for all scheduled visits.
5. In the Investigator's opinion, subject is able to understand the nature of the study and any risks involved in participation, and willing to cooperate and comply with the protocol restrictions and requirements (including travel).
6. Female subjects who are non-lactating and have a negative urine pregnancy test at baseline visit prior to receiving the first dose of study drug.
7. Female subjects of childbearing potential and male subjects with partner of child-bearing potential currently using/willing to use 2 effective methods of contraception including barrier method as described in the protocol.

Exclusion Criteria:

1. History or presence of photodermatoses other than EPP or XLP.
2. Subjects who are unwilling or unable to go outside during daylight hours most days (e.g., between 1 hour post sunrise and 1 hour pre-sunset) during the study.
3. Presence of clinically significant hepatobiliary disease based on LFT values at Screening.
4. Subjects with AST, ALT, ALP ≥3.0 × upper limit of normal (ULN) or total bilirubin >1.5 × ULN at Screening.
5. Subjects with or having a history (in the last 2 years) of excessive alcohol intake in the opinion of the Investigator.
6. History of melanoma.
7. Presence of melanoma and/or lesions suspicious for melanoma at Screening.
8. History of familial melanoma (defined as having 2 or more first-degree relatives, such as parents, sibling and/or child).
9. Presence of squamous cell carcinoma, basal cell carcinoma, or other malignant skin lesions.

   Any suspicious lesions or nevi will be evaluated. If the suspicious lesion or nevi cannot be resolved through biopsy or excision, the subject will be excluded from the study.
10. History or presence of psychiatric disease judged to be clinically significant by the Investigator and which may interfere with the study evaluation and/or safety of the subjects.
11. Presence of clinically significant acute or chronic renal disease based upon the subject's medical records including hemodialysis; an estimated glomerular filtration rate (eGFR) <60 mL/min as calculated by the Chronic Kidney Disease-Epidemiology Collaboration (CKDEPI) creatinine equation (2009) for adults and by the Schwartz creatinine equation for adolescents (2009). Modification of Diet in Renal Disease (MDRD) can be used for adults per local recommendations.
12. Presence of any clinically significant disease or laboratory abnormality which, in the opinion of the Investigator, can interfere with the study objectives and/or safety of the subjects.
13. Female subjects who are pregnant, lactating, or intending to become pregnant during the study.
14. Treatment with phototherapy within 3 months before Randomization (Visit 2).
15. Treatment with afamelanotide within 3 months before Randomization (Visit 2).
16. Treatment with cimetidine within 4 weeks before Randomization (Visit 2).
17. Treatment with antioxidant agents within 4 weeks before Randomization (Visit 2), at doses which, in the opinion of the Investigator, may affect study endpoints (including but not limited to beta-carotene, cysteine, pyridoxine).
18. Chronic treatment with any scheduled analgesic agents including, but not limited to, opioids and opioid derivatives such as morphine, hydrocodone, oxycodone, fentanyl, or their combination with other unscheduled analgesics or non-steroidal anti-inflammatory drug (Percocet and Vicodin-like prescription drugs) within 4 weeks before Randomization (Visit 2).

    Acute use of scheduled narcotics greater than 3 months prior to randomization, OTCs, such as NSAIDs or aspirin for analgesia, or prior temporary use of scheduled agents within 3 months of screening are not excluded.
19. Treatment with any drugs or supplements which, in the opinion of the Investigator, can interfere with the objectives of the study or safety of the subjects.
20. Previous exposure to MT-7117 (this does not include placebo treated subjects).
21. Previous treatment with any investigational agent within 12 weeks before Screening OR 5 half-lives of the investigational product (whichever is longer).

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-12-14 (Actual); Study Completion 2022-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Head of Medical Science, Study Director — Tanabe Pharma America, Inc.
Locations (31):
- United States (10):
  - Marvel Clinical Research, LLC, Huntington Beach, California
  - University Of Miami School Of Medicine, Center For Liver Diseases, Miami, Florida
  - MetroBoston Clinical Partners, LLC, Brighton, Massachusetts
  - Kansas City Research Institute, Kansas City, Missouri
  - Icahn School of Medicine at Mount Sinai (ISMMS) - The Mount Sinai Hospital (MSH), New York, New York
  - Wake Forest University Baptist Health, Winston-Salem, North Carolina
  - Remington-Davis Clinical Research, Columbus, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - The University of Texas Medical Branch (UTMB), Galveston, Texas
  - University of Washington-Seattle Cancer Care Alliance, Seattle, Washington
- Australia (2):
  - The Wesley Hospital, Brisbane, Queensland
  - Royal Melbourne Hospital (RMH), Melbourne, Victoria
- University of Alberta, Edmonton, Alberta, Canada
- Germany (2):
  - Westfaelische Wilhelms-Universitaet Muenster, Münster, Northrhein Westalien
  - Charite - Universitaetsmedizin Berlin, Berlin
- Italy (4):
  - Azienda Ospedaliera Spedali Civili di Brescia-Universita degli Studi Di Brescia, Brescia
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico di Milano, Milan
  - U.O.C. Medicina Interna Azienda ospedaliero Universitaria Policlinico di Modena, Modena
  - I.F.O Hospital Centro Porfirie e Malattie Rare, Rome
- Japan (6):
  - Kobe University Hospital, Kobe, Hyōgo
  - Sophia Dermatology Clinic, Kanazawa, Ishikawa-ken
  - Investigator site, Sayama, Osaka
  - Osaka Medical College Hospital, Takatsuki, Osaka
  - Tokyo Saiseikai Central Hospital, Minato-ku, Tokyo
  - Toyama University Hospital, Sugitani, Toyama
- Haukeland University Hospital, Bergen, Norway
- Spain (2):
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
- Karolinska University Hospital, Stockholm, Sweden
- United Kingdom (2):
  - University of Manchester, Salford, Manchester
  - Evelina London Children's Hospital - Guy's & St Thomas' NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ogasawara A, Ide R, Inoue S, Tsuda M, Teng R. Assessment of Potential Drug-Drug Interactions for Novel Oral Melanocortin-1 Receptor Agonist Dersimelagon. Pharmacol Res Perspect. 2025 Feb;13(1):e70069. doi: 10.1002/prp2.70069. PMID 39887900

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Subjects who were randomized to receive matching oral tablet of placebo once a day in Double-Blind treatment
- MT-7117 Low Dose: Subjects who were randomized to receive oral tablet of MT-7117 Low Dose once a day in Double-Blind Treatment and Double-Blind Extension
- MT-7117 High Dose: Subjects who were randomized to receive oral tablet of MT-7117 High Dose once a day in Double-Blind Treatment and Double-Blind Extension
- Placebo -> MT-7117 Low Dose: Subjects who received placebo in Double-Blind Treatment, and after that received MT-7117 low dose in Double-Blind Extension
- Placebo -> MT-7117 High Dose: Subjects who received placebo in Double-Blind Treatment, and after that received MT-7117 high dose in Double-Blind Extension
Period: 26 Weeks Double-Blind Treatment (DBT)
Arm/Group | Placebo | MT-7117 Low Dose | MT-7117 High Dose | Placebo -> MT-7117 Low Dose | Placebo -> MT-7117 High Dose
Started | 61 | 63 | 60 | 0 | 0
Completed | 57 | 60 | 58 | 0 | 0
Not Completed | 4 | 3 | 2 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 2 | 2 | 0 | 0
Period: 26 Weeks Double-Blind Extension (DBE)
Arm/Group | Placebo | MT-7117 Low Dose | MT-7117 High Dose | Placebo -> MT-7117 Low Dose | Placebo -> MT-7117 High Dose
Started | 0 (Of 57 participants randomized to placebo in 26 weeks double-blind period, 28 were re-randomized to MT-7117 low dose, and 28 were re-randomized to MT-7117 high dose. 1 participant did not take the offer to participate in period 2) | 56 (4 participants did not take the offer to participate in period 2) | 55 (3 participants did not take the offer to participate in period 2) | 28 (Of 57 participants who were randomized to placebo in period 1, 28 participants were allocated to MT-7117 low dose in period 2) | 28 (Of 57 participants who were randomized to placebo in period 1, 28 participants were allocated to MT-7117 high dose in period 2)
Completed | 0 | 55 | 52 | 27 | 28
Not Completed | 0 | 1 | 3 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | MT-7117 Low Dose | MT-7117 High Dose | Total
Number analyzed (Participants) | 61 | 63 | 60 | 184
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12 | 13 | 12 | 37
  Between 18 and 65 years | 47 | 45 | 46 | 138
  >=65 years | 2 | 5 | 2 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 30 | 33 | 93
  Male | 31 | 33 | 27 | 91
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 7 | 2 | 16
  Not Hispanic or Latino | 53 | 52 | 58 | 163
  Unknown or Not Reported | 1 | 4 | 0 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 9 | 1 | 2 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 0 | 0 | 0 | 0
  White | 52 | 60 | 55 | 167
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Average Daily Sunlight Exposure Time (Minutes) to First Prodromal Symptom (Burning, Tingling, Itching, or Stinging) Associated With Sunlight Exposure Between 1 Hour Post Sunrise and 1 Hour Pre-sunset at Week 26 (Visit 7)
Time Frame: From 1 hour post-sunrise to 1 hour pre-sunset at Week 26 (Visit 7)
Population: Included all randomized subjects who received at least 1 dose of study medication with Baseline and post randomization- sunlight exposure diary assessments during the double-blind treatment period.
Measure: Least Squares Mean (Standard Error); unit: minute
Groups:
- DBT ITT1 Placebo: Oral tablet of placebo once a day in DBT
- DBT ITT1 MT- 7117 Low Dose: Oral tablet of MT-7117 Low Dose once a day in DBT
- DBT ITT1 MT- 7117 High Dose: Oral tablet of MT-7117 High Dose once a day in DBT
Arm/Group | DBT ITT1 Placebo | DBT ITT1 MT- 7117 Low Dose | DBT ITT1 MT- 7117 High Dose
Number analyzed (Participants) | 60 | 63 | 60
minute | 20.59 (10.29) | 30.39 (10.04) | 43.29 (10.13)
Statistical Analysis 1: Comparison: DBT ITT1 Placebo vs DBT ITT1 MT- 7117 Low Dose; Change from BL at Week 26 (DBT EOT) - lower dose; Test type: Superiority; p = 0.496, Mixed-effect model for repeated measures; Least Square Mean Difference vs Placebo = 9.8, 95% CI 2-sided [-18.52 to 38.12], Standard Error of Mean 14.35
Statistical Analysis 2: Comparison: DBT ITT1 Placebo vs DBT ITT1 MT- 7117 High Dose; Change from BL at Week 26 (DBT EOT) - higher dose; Test type: Superiority; p = 0.116, Mixed-effect model for repeated measures; Least Square Mean Difference vs Placebo = 22.7, 95% CI 2-sided [-5.68 to 51.09], Standard Error of Mean 14.38

2. Secondary Outcome: Patient Global Impression of Change (PGIC) at Week 26
Description: PGIC: Scale from 1 to 7, where 7 is worse.
Time Frame: Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: point
Arm/Group | DBT ITT1 Placebo | DBT ITT1 MT- 7117 Low Dose | DBT ITT1 MT- 7117 High Dose
Number analyzed (Participants) | 56 | 59 | 56
point | 3.25 (1.14) | 2.41 (0.14) | 1.82 (0.14)
Statistical Analysis 1: Comparison: DBT ITT1 Placebo vs DBT ITT1 MT- 7117 Low Dose; Test type: Superiority; p < 0.001, Mixed-effect model for repeated measures; Least Square Mean Difference vs Placebo = -0.84, 95% CI 2-sided [-1.23 to -0.44], Standard Error of Mean 0.2
Statistical Analysis 2: Comparison: DBT ITT1 Placebo vs DBT ITT1 MT- 7117 High Dose; Test type: Superiority; p < 0.001, Mixed-effect model for repeated measures; Least Square Mean Difference vs Placebo = -1.43, 95% CI 2-sided [-1.83 to -1.03], Standard Error of Mean 0.2

3. Secondary Outcome: Total Number of Sunlight-induced Pain Events Defined as Prodrome Symptoms (Burning, Tingling, Itching, or Stinging) With Pain Rating of 1-10 on the Likert Scale During the 26-week Double-blind Treatment Period.
Description: The Likert scale used ranges from 0 to 10, where 0 indicates the lowest pain rating and 10 indicates the highest pain rating. Likewise, 0 indicates to best outcome and 10 indicates the worst outcome. The sum of the number of pain events with pain rating of 1 to 10 for the day is used as the number of sunlight-induced pain events in the day. The sum of the number of the pain events with pain rating of 1 to 10 in each day during the 26-week Double-blind Treatment Period is calculated as this endpoint.
Time Frame: During the 26-week double-blind treatment period
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: events
Arm/Group | DBT ITT1 Placebo | DBT ITT1 MT- 7117 Low Dose | DBT ITT1 MT- 7117 High Dose
Number analyzed (Participants) | 60 | 63 | 60
events | 23.9 (30.93) | 15.87 (22.05) | 13.78 (18.7)
Statistical Analysis 1: Comparison: DBT ITT1 Placebo vs DBT ITT1 MT- 7117 Low Dose; Test type: Superiority — Negative binomial regression model with log link was used; p = 0.199, Refer to comments below:; Negative binomial regression model with log link was used for other method; Incident rate ratio = 0.76, 95% CI 2-sided [0.49 to 1.16]
Statistical Analysis 2: Comparison: DBT ITT1 Placebo vs DBT ITT1 MT- 7117 High Dose; Test type: Superiority — Negative binomial regression model with log link was used; p = 0.006, Refer to comments below:; Negative binomial regression model with log link was used for other method; Incident rate ratio = 0.55, 95% CI 2-sided [0.36 to 0.84]

4. Secondary Outcome: Change From Baseline for Total Score in the Domain of Pain Intensity in the PROMIS-57 at Week 26
Description: Pain intensity: 0 to 10, where 10 is worst pain imaginable.
Time Frame: Baseline (Week 0) and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: total score
Arm/Group | DBT ITT1 Placebo | DBT ITT1 MT- 7117 Low Dose | DBT ITT1 MT- 7117 High Dose
Number analyzed (Participants) | 49 | 59 | 56
total score | -1.42 (0.18) | -1.56 (0.16) | -1.65 (0.17)
Statistical Analysis 1: Comparison: DBT ITT1 Placebo vs DBT ITT1 MT- 7117 Low Dose; Test type: Superiority; p = 0.55, mixed-effect model for repeated measures; Least Square Mean Difference vs Placebo = -0.15, 95% CI 2-sided [-0.62 to 0.33], Standard Error of Mean 0.24
Statistical Analysis 2: Comparison: DBT ITT1 Placebo vs DBT ITT1 MT- 7117 High Dose; Test type: Superiority; p = 0.343, mixed-effect model for repeated measures; Least Square Mean Difference vs Placebo = -0.23, 95% CI 2-sided [-0.72 to 0.25], Standard Error of Mean 0.25

5. Secondary Outcome: The Percentage of Subjects Who Are Responders
Description: The percentage of subjects who are responders based on average daily sunlight exposure time to first prodromal symptom associated with sunlight exposure between 1 hour post-sunrise and 1 hour presunset defined by within-subject meaningful change of 66 minutes increase from baseline to Week 26
Time Frame: Week 26
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | DBT ITT1 Placebo | DBT ITT1 MT- 7117 Low Dose | DBT ITT1 MT- 7117 High Dose
Number analyzed (Participants) | 60 | 63 | 60
percentage of participants | 12 | 11 | 16
Statistical Analysis 1: Comparison: DBT ITT1 Placebo vs DBT ITT1 MT- 7117 Low Dose; Test type: Superiority; p = 0.642, Regression, Logistic; Odds Ratio (OR) = 0.805, 95% CI 2-sided [0.323 to 2.007]
Statistical Analysis 2: Comparison: DBT ITT1 Placebo vs DBT ITT1 MT- 7117 High Dose; Test type: Superiority; p = 0.431, Regression, Logistic; Odds Ratio (OR) = 1.412, 95% CI 2-sided [0.598 to 3.336]

6. Secondary Outcome: Change From Baseline for Total Score in the Domain of Physical Function in the PROMIS-57 at Week 26
Description: Physical function: 1-5, where 5 is without any difficulty.
Time Frame: Baseline (Week 0) and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: total score
Arm/Group | DBT ITT1 Placebo | DBT ITT1 MT- 7117 Low Dose | DBT ITT1 MT- 7117 High Dose
Number analyzed (Participants) | 49 | 59 | 56
total score | 0.67 (0.36) | 1.54 (0.32) | 1.22 (0.33)
Statistical Analysis 1: Comparison: DBT ITT1 Placebo vs DBT ITT1 MT- 7117 Low Dose; Test type: Superiority; p = 0.072, mixed-effect model for repeated measures; Least Square Mean Difference vs Placebo = 0.87, 95% CI 2-sided [-0.08 to 1.82], Standard Error of Mean 0.48
Statistical Analysis 2: Comparison: DBT ITT1 Placebo vs DBT ITT1 MT- 7117 High Dose; Test type: Superiority; p = 0.252, mixed-effect model for repeated measures; Least Square Mean Difference vs Placebo = 0.56, 95% CI 2-sided [-0.4 to 1.51], Standard Error of Mean 0.48

ADVERSE EVENTS:
Time Frame: through study completion, an average of 58 weeks
Description: Total Number At Risk of Adverse event is the number of patients who enrolled in DBT or DBE period and who received at least 1 dose of study medication during the period. For "DBE: MT-7117 high dose", 55 patients were enrolled in DBE period and 54 patients received at least 1 dose of study medication during DBE period. Therefore, 54 patients are the Total Number At Risk for "DBE: MT-7117 high dose".
Groups:
- DBT: Placebo: Subjects who were randomized to receive matching oral tablet of placebo once a day in Double-Blind Treatment
- DBT: MT-7117 Low Dose: Subjects who were randomized to receive oral tablet of MT-7117 Low Dose once a day in Double-Blind Treatment
- DBT: MT-7117 High Dose: Subjects who were randomized to receive oral tablet of MT-7117 High Dose once a day in Double-Blind Treatment
- DBE: MT-7117 Low Dose Switched From Placebo: Subjects who received MT-7117 low dose in Double-Blind Extension The subjects were switched from Placebo for Double-Blind Extension.
- DBE: MT-7117 High Dose Switched From Placebo: Subjects who received MT-7117 high dose in Double-Blind Extension. The subjects were switched from Placebo for Double-Blind Extension.
- DBE: MT-7117 Low Dose: Subjects who received oral tablet of MT-7117 Low Dose once a day in Double-Blind Extension
- DBE: MT-7117 High Dose: Subjects who were received oral tablet of MT-7117 High Dose once a day in Double-Blind Extension
Arm/Group | DBT: Placebo | DBT: MT-7117 Low Dose | DBT: MT-7117 High Dose | DBE: MT-7117 Low Dose Switched From Placebo | DBE: MT-7117 High Dose Switched From Placebo | DBE: MT-7117 Low Dose | DBE: MT-7117 High Dose
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/63 | 1/60 | 0/28 | 0/28 | 0/56 | 0/54
Serious Adverse Events (participants affected / at risk) | 0/61 | 2/63 | 2/60 | 2/28 | 1/28 | 1/56 | 2/54
Other Adverse Events (participants affected / at risk) | 30/61 | 35/63 | 40/60 | 19/28 | 18/28 | 24/56 | 21/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DBT: Placebo (N=61) | DBT: MT-7117 Low Dose (N=63) | DBT: MT-7117 High Dose (N=60) | DBE: MT-7117 Low Dose Switched From Placebo (N=28) | DBE: MT-7117 High Dose Switched From Placebo (N=28) | DBE: MT-7117 Low Dose (N=56) | DBE: MT-7117 High Dose (N=54)
Myocarditis (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Porphyria non-acute (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Meningitis viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DBT: Placebo (N=61) | DBT: MT-7117 Low Dose (N=63) | DBT: MT-7117 High Dose (N=60) | DBE: MT-7117 Low Dose Switched From Placebo (N=28) | DBE: MT-7117 High Dose Switched From Placebo (N=28) | DBE: MT-7117 Low Dose (N=56) | DBE: MT-7117 High Dose (N=54)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Porphyria non-acute (Congenital, familial and genetic disorders) | 5 | 1 | 1 | 2 | 1 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 4 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 5 | 8 | 0 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 4 | 4 | 17 | 1 | 5 | 1 | 2
Cyst (General disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Fatigue (General disorders) | 4 | 3 | 3 | 0 | 1 | 2 | 1
COVID-19 (Infections and infestations) | 2 | 5 | 1 | 7 | 8 | 11 | 10
Nasopharyngitis (Infections and infestations) | 1 | 1 | 1 | 2 | 0 | 4 | 3
Upper respiratory tract infection (Infections and infestations) | 5 | 1 | 2 | 1 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 1 | 2 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 3 | 0 | 2 | 0 | 1 | 2
Aspartate aminotransferase increased (Investigations) | 1 | 4 | 0 | 3 | 1 | 1 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 1 | 3 | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 5 | 3 | 1 | 2 | 1 | 1 | 0
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 3 | 1
Vitamin D decreased (Investigations) | 1 | 0 | 0 | 2 | 0 | 1 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 4 | 2
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0 | 3 | 1 | 3 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 2 | 0 | 0 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 6 | 8 | 4 | 3 | 3 | 2
Headache (Nervous system disorders) | 3 | 8 | 9 | 2 | 3 | 2 | 2
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 3 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0
Ephelides (Skin and subcutaneous tissue disorders) | 1 | 3 | 4 | 0 | 0 | 0 | 0
Nail pigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 2 | 0 | 0 | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 6 | 1 | 2 | 1 | 2 | 0 | 2
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 5 | 6 | 0 | 1 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 3 | 8 | 2 | 3 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 2 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2021-08-09): https://cdn.clinicaltrials.gov/large-docs/89/NCT04402489/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-16): https://cdn.clinicaltrials.gov/large-docs/89/NCT04402489/SAP_001.pdf